CLINICAL TRIAL: NCT06057662
Title: Effect of Personalized Comprehensive Diabetes Support Among Families of Children With Newly Diagnosed Type 1 Diabetes
Brief Title: Personalized Comprehensive Diabetes Support for Children With Newly Diagnosed Type 1 Diabetes
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2059749
Record Dates: First submitted 2023-08-08; First posted 2023-09-28 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): personalized comprehensive diabetes support for 6 months following type 1 diabetes diagnosis
  Interventions: Other: personalized comprehensive diabetes support
- Control (No Intervention)

INTERVENTIONS:
Other: personalized comprehensive diabetes support — personalized comprehensive diabetes support
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to learn if access to a diabetes coach improves quality of life (QOL) for families of children with newly diagnosed type 1 diabetes. The main questions it aims to answer are:

1. Determine if there are beneficial effects on diabetes-related QOL at the end of the 6-month intervention.
2. Determine if potential beneficial effects persist beyond completion of the support intervention, as measured by diabetes-related QOL at 12 months and 24 months following diagnosis

Participants assigned to the intervention group will have access to a diabetes coach for 6 months following type 1 diabetes diagnosis. They will be compared to participants who are assigned to the control group and are receiving usual care.

ELIGIBILITY:
Inclusion Criteria:

* Families of children 16 years of age or younger with a new diagnosis
* Stable living situation such that the same caregivers are anticipated to be caring for the child during the full 2-year study duration.

Exclusion Criteria:

* Families of children older than 16 years
* Children from non-English speaking families

Ages: 0 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Diabetes Distress Scale | 24 months
  The Distress Scale (DDS) uses a 6-point Likert scale to quantify diabetes-related stress. Scores can range from 0 to 72. A higher score indicates higher distress.
Problem Areas in Diabetes (PAID) | 24 months
  The Problem Areas in Diabetes (PAID) uses a 6-point Likert scale to quantify diabetes-related stress. Scores can range from 0 to 100. A higher score indicates higher distress.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No